CLINICAL TRIAL: NCT06525909
Title: A Real-world Study of Staging and Grading of Clinical Immune Status in Chronic Hepatitis B
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Other Study IDs: OCEAN cure 06 study
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Untreated group: The untreated patients who met the staging subgroups of the Chinese Guidelines for the Prevention and Control of Chronic Hepatitis B, 2022 edition or lost HBsAg spontaneously.
- NA treatment group: The patients who achieved HBV DNA suppression by NA.

SUMMARY:
This is a prospective, multicentre observational study of Chronic Hepatitis B （CHB）in different clinical stages. We intend to compare the immune status of various types of CHB patients, and we propose to establish a staging and grading criteria for the immune exhaustion status of patients with CHB.

DETAILED DESCRIPTION:
Two groups were included in this study: untreated patients who met the staging subgroups according to Chinese Guidelines for the Prevention and Control of Chronic Hepatitis B, 2022 edition or HBsAg negativity（Group 1). The another is those who achieved HBV DNA suppression by NA（Group 2）. Patients in Group 1 will be followed up once every six months, and in group 2 will be followed up once every three months. And patients treated or not treated will be followed up in the study. The treatment with NA or combined with interferon will be decided by the consensus of doctors and patients. This study does not intervene the treatment, but will register the clinical indicators. We follow up the patients at each follow-up time point, record the subjects' clinical indicators at each visit and obtained serum and PBMC specimens for further immune study after the consents of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CHB who were older than 18 years old and younger than 50 years old with HBsAg positivity more than 6 months;
2. Group 1 untreated group fulfils any one of the four natural history types of the Chinese Guidelines for the Prevention and Control of Chronic Hepatitis B, 2022.
3. Group 2 nucleos(t)ide-treated CHB patients are required to have sustained control of their HBV DNA (<100 IU/ml).

Exclusion Criteria:

1. Pregnancy status;
2. Has been diagnosed with compensated/lost compensated cirrhosis, hepatocellular carcinoma by imaging or other indicators;
3. Combined HAV, HCV, HEV infection, schistosomal liver disease, drug-induced liver injury, autoimmune hepatitis, alcoholic liver disease, severe fatty liver, HIV infection;
4. Being on immunosuppressants or immunomodulators or hormonal drugs or biological agents, etc;
5. previous history of oncology, organ transplantation, etc., history of alcoholism (>30 g/d for men, >20 g/d for women);
6. Inadequate follow-up time and inadequate clinical/laboratory information;
7. Combined heart, brain, kidney, lung and other organ insufficiency or combined endocrine and haematological system and other major diseases;
8. Comorbid serious psychiatric diseases including severe anxiety or depression;
9. Unwilling to participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the patients with Chronic Hepatitis B
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
A preliminary exploration of staging and grading criteria for the state of immune | week 200
  The clinical characteristics, viral load and immune cells frequency (CD4+ or CD8+ T cells, etc) of CHB in different clinical stages will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Doctor, Principal Investigator — Department of infectious Diseases, Tongji Hospital
Locations (5):
- China (5):
  - Tongji Hospital, Wuhan, Hubei
  - Beijing YouAn Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Southwest Hospital, Chongqing
  - Jiangsu Province Hospital, Nanjing

IPD SHARING:
Plan to Share IPD: Undecided